CLINICAL TRIAL: NCT04299048
Title: A PHASE 1B, 12-WEEK, OPEN-LABEL STUDY TO ASSESS THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND PHARMACODYNAMICS FOLLOWING REPEATED SUBCUTANEOUS ADMINISTRATIONS OF PF-06946860 IN PATIENTS WITH CANCER AND CACHEXIA
Brief Title: Study to Assess the Safety and Tolerability of Repeated Doses of an Investigational New Drug in Patients With Cancer and Cachexia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C3651009
Record Dates: First submitted 2020-02-19; First posted 2020-03-06 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-03

CONDITIONS: Cachexia; Non-Small-Cell Lung Cancer; Pancreatic Cancer; Colorectal Cancer
Keywords: cachexia, non-small cell lung cancer, pancreatic cancer; colorectal cancer, weight loss, anorexia, muscle loss, fatigue
MeSH Terms: conditions — Cachexia; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Colorectal Neoplasms; Weight Loss; Anorexia; Muscular Atrophy; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06946860 (Experimental): subcutaneous injection
  Interventions: Drug: PF-06946860

INTERVENTIONS:
Drug: PF-06946860 — subcutaneous injection

SUMMARY:
Study to assess the safety and tolerability of repeated doses of an investigational new drug in patients with cancer and cachexia.

DETAILED DESCRIPTION:
This 12-week open-label study will explore how PF-06946860 is tolerated, the effects of the study drug, the best dose for treatment and how participants with non-small cell lung, pancreatic or colorectal cancer and cachexia feel after receiving repeated subcutaneous dosing. During the 12-week treatment period, study drug will be administered subcutaneously every 3 weeks for a total of 5 doses. There is a 12-week follow-up period following the last dose of study drug. Additional assessments include:

* body weight measurements
* blood pressure and heart rate measurements
* Lumbar Skeletal Muscle Index (LSMI) by CT scan
* Blood samples:

  * to evaluate safety,
  * to measure the amount of the study drug in the blood,
  * to evaluate if the study drug causes an immune response,
  * to examine the effects of the study drug on levels of a specific cytokine,
  * and for exploratory samples for bio banking.
* Measure the impact of the study drug on appetite, nausea, vomiting, fatigue, physical function, and health-related quality of life with questionnaires.
* Measure the impact of study drug on physical activity using wearable digital sensors.
* To evaluate the effect of study drug on ability to complete anti-tumor treatment and survival in participants with cancer and cachexia.
* To evaluate tumor size.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologic or cytologic diagnosis of advanced metastatic NSCLC, advanced/unresectable pancreatic cancer, or metastatic colorectal cancer.
* Cachexia, defined by BMI <20 kg/m2 with involuntary weight loss of >2% within 6 months prior to screening or Involuntary weight loss of >5% within 6 months prior to screening irrespective of BMI or If medical record documentation is unavailable, patient's report will suffice to estimate involuntary body weight loss.;
* Will receive the following for non-small cell lung cancer:

  * a platinum + pemetrexed ± pembrolizumab or
  * a platinum + nab paclitaxel or paclitaxel ± pembrolizumab or
  * pembrolizumab alone
* Will receive the following for pancreatic cancer:

  * FOLFIRINOX or
  * Nab-Paclitaxel + Gemcitabine
  * Gemcitabine
* Will receive the following for colorectal cancer:

  * FOLFOX +/- Biologic (Bevacizumab or Cetuximab/Panitumumab) or
  * FOLFIRI +/- Biologic (Bevacizumab or Cetuximab/Panitumumab) or
  * FOLFOXIRI +/- Biologic (Bevacizumab or Cetuximab/Panitumumab) or
  * Pembrolizumab for MSI-H • Will be entering the study at the first or second cycle of their current course of anti-cancer treatment/ therapy.
* Adequate renal and liver function.
* Signed informed consent.

Exclusion Criteria:

* All other forms of cancers not specified above unless currently considered cured (>5 years without evidence of recurrence).
* Planned radiation therapy as part of the primary anti-tumor therapy regimen. However, localized radiation therapy for symptomatic relief is permitted
* Cachexia caused by other reasons: Severe COPD requiring use of home O2, heart failure or AIDS.
* known symptomatic brain metastases requiring steroids.
* Active hepatitis B or C virus.
* Confirmed positive HIV test.
* Current active reversible causes of decreased food intake.
* Receiving tube feedings or parenteral nutrition at Screening.
* Elevated blood pressure that cannot be controlled by medications.
* Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - SCL Health Cancer Centers of Colorado - St. Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Lutheran Medical Center, Wheat Ridge, Colorado
  - Tallahassee Memorial Healthcare Cancer Center, Tallahassee, Florida
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - New England Cancer Specialists, Scarborough, Maine
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - American Oncology Partners of Maryland, PA, Germantown, Maryland
  - Duke Cancer Center, Durham, North Carolina
  - VA Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3651009

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 20 participants were screened for eligibility, of which 11 participants were enrolled into the study. A total of 10 participants were treated.
Groups:
- PF-06946860 Q3W: During the 12-week treatment period, participants receive a total of 5 subcutaneously (SC) doses of PF-06946860 every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | PF-06946860 Q3W
Started | 11
Treated | 10
Completed | 7
Not Completed | 4
Not completed — Death | 1
Not completed — Global deterioration of health status | 2
Not completed — Enrolled and not treated | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis was performed on treated participants.
Groups:
- PF-06946860 Q3W: During the 12-week treatment period, participants receive a total of 5 SC doses of PF-06946860 Q3W.
Arm/Group | PF-06946860 Q3W
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Body Mass Index [Median (Full Range); unit: kg/m^2] | 22.88 [17.31 to 30.87]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) was defined as an AE: 1. resulting in death, 2. was life-threatening, 3. required inpatient hospitalization or prolongation of existing hospitalization, 4. resulted in persistent disability, 5. was a congenital anomaly/birth defect, or considered to be an important medical event. An AE was considered an TEAE if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the last dose plus the lag time were flagged as TEAEs.
Time Frame: From Day 1 up to Week 24
Population: The safety analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06946860 Q3W
Number analyzed (Participants) | 10
Participants
  AEs | 10
  SAEs | 4

2. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Participants with laboratory test abnormalities (without regard to baseline abnormality) that met pre-specified criteria included Hemoglobin< 0.8x lower limit of normal (LLN); Hematocrit< 0.8x LLN; Erythrocytes (Ery.)< 0.8x LLN; Ery. Mean Corpuscular Volume< 0.9x LLN; Leukocytes< 0.6x LLN; Lymphocytes< 0.8x LLN; Bilirubin> 1.5x upper limit of normal (ULN); Aspartate Aminotransferase> 3.0x ULN; Alkaline Phosphatase> 3.0x ULN; Protein< 0.8x LLN; Sodium< 0.95x LLN; Chloride< 0.9x LLN; Calcium< 0.9x LLN; Bicarbonate< 0.9x LLN; Glucose> 1.5x ULN; C Reactive Protein> 1.1x ULN; for urinalysis, Urine Glucose ≥1, Ketones ≥1, Urine Protein ≥1, Urine Hemoglobin ≥1, Urobilinogen ≥1, Nitrite ≥1, and Leukocyte ≥1 Esterase ≥1; Hyaline Casts >1/LPF.
Time Frame: From Day 1 up to Week 24
Population: Overall number of participants analyzed included participants with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06946860 Q3W
Number analyzed (Participants) | 8
Participants
  Hemoglobin (g/dL)< 0.8x LLN | 2
  Hematocrit (%)< 0.8x LLN | 2
  Erythrocytes (10^6/mm^3)< 0.8x LLN | 2
  Ery. Mean Corpuscular Volume (um^3)< 0.9x LLN | 1
  Leukocytes (10^3/mm^3)< 0.6x LLN | 2
  Lymphocytes (10^3/mm^3)< 0.8x LLN | 3
  Bilirubin (mg/dL)> 1.5x ULN | 1
  Aspartate Aminotransferase (U/L)> 3.0x ULN | 1
  Alkaline Phosphatase (U/L)> 3.0x ULN | 2
  Protein (g/dL)< 0.8x LLN | 1
  Sodium (mEq/L)< 0.95x LLN | 1
  Chloride (mEq/L)< 0.9x LLN | 1
  Calcium (mg/dL)< 0.9x LLN | 1
  Bicarbonate (mEq/L)< 0.9x LLN | 2
  Glucose (mg/dL)> 1.5x ULN | 4
  C Reactive Protein (mg/dL)> 1.1x ULN | 5
  URINE Glucose ≥1 | 3
  Ketones ≥1 | 1
  URINE Protein ≥1 | 1
  URINE Hemoglobin ≥1 | 2
  Urobilinogen ≥1 | 1
  Nitrite ≥1 | 1
  Leukocyte Esterase ≥1 | 2
  Hyaline Casts >1/LPF: number analyzed (Participants) | 3
  Hyaline Casts >1/LPF | 2

3. Primary Outcome: Number of Participants With Post-Baseline Vital Signs Abnormalities
Description: Vital signs (pulse rate, systolic and diastolic blood pressure) were obtained with participant in the supine position. The pre-specified categorical analysis criteria in vital signs, were supine systolic blood pressure (SBP) <90 millimeters of mercury (mmHg), supine SBP increase/decrease from baseline ≥30 mmHg; supine diastolic blood pressure (DBP) <50 mmHg, supine DBP increase/decrease from baseline ≥20 mmHg; supine pulse rate <40 beats per minute (bpm) or >120 bpm.
Time Frame: From Day 1 up to Week 24
Population: Overall number of participants analyzed included participants evaluated against pre-defined criteria for vital signs.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06946860 Q3W
Number analyzed (Participants) | 9
Participants
  Supine SBP - Value <90 mmHg | 0
  Supine SBP - Change ≥ 30 mmHg Increase | 2
  Supine SBP - Change ≥ 30 mmHg Decrease | 0
  Supine DBP - Value <50 mmHg | 0
  Supine DBP - Change ≥ 20 mmHg Increase | 1
  Supine DBP - Change ≥ 20 mmHg Decrease | 0
  Supine Pulse Rate - Value <40 bpm | 0
  Supine Pulse Rate - Value >120 bpm | 0

4. Primary Outcome: Number of Participants With Post-Baseline Electrocardiogram (ECG) Abnormalities
Description: ECG data (PR interval, QRS interval, QT interval, and QTcF) were obtained with participant in the supine position. The pre-specified categorical analysis criteria in ECG, were PR interval: value ≥300 milliseconds (msec), percentage change ≥25/50%; QRS interval: value ≥140 msec, percentage change ≥50%; QT interval: value ≥500 msec; QTcF interval: 470< value ≤480 msec, 480< value ≤500 msec, value >500 msec, and 30< change ≤60 msec, change >60 msec.
Time Frame: From Day 1 up to Week 24
Population: Overall number of participants analyzed included participants evaluated against pre-defined criteria for ECGs.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06946860 Q3W
Number analyzed (Participants) | 8
Participants
  Supine PR Interval - Value ≥300 msec | 0
  Supine PR Interval - %Chg ≥25/50% | 0
  Supine QRS Interval - Value ≥140 msec | 0
  Supine QRS Interval - %Chg ≥50% | 0
  Supine QT Interval - Value ≥500 msec | 0
  Supine QTcF - 470<Value≤480 msec | 0
  Supine QTcF - 480<Value≤500 msec | 0
  Supine QTcF - Value>500 msec | 0
  Supine QTcF - 30<Chg≤60 msec | 2
  Supine QTcF - Chg>60 msec | 0

5. Secondary Outcome: Serum Unbound Trough Concentrations (Ctrough) of PF-06946860
Description: Ctrough was defined as the samples measured pre-dose at Weeks 3, 6, 9 and 12, and at Week 15. Serum unbound Ctrough was summarized by time and treatment group.
Time Frame: Pre-dose at Weeks 3, 6, 9 and 12, and at Week 15
Population: The analysis set included all randomized participants who received a dose of PF-06946860 and in whom at least 1 serum concentration value was reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06946860 Q3W
Number analyzed (Participants) | 8
ng/mL
  Week 3 | 4.041 (1.28*10^19)
  Week 6 | 1690 (593)
  Week 9 | 610.9 (7.79*10^10)
  Week 12 | 4383 (142)
  Week 15: number analyzed (Participants) | 7
  Week 15 | 560.5 (2.15*10^12)

6. Secondary Outcome: Serum Total Ctrough of PF-06946860
Description: Ctrough was defined as the samples measured pre-dose at Weeks 3, 6, 9 and 12, and at Week 15. Serum total Ctrough was summarized by time and treatment group.
Time Frame: Pre-dose at Weeks 3, 6, 9 and 12, and at Week 15
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06946860 Q3W
Number analyzed (Participants) | 8
ng/mL
  Week 3 | 10050 (19)
  Week 6 | 17010 (16)
  Week 9 | 20740 (24)
  Week 12 | 21310 (32)
  Week 15: number analyzed (Participants) | 7
  Week 15 | 25450 (31)

ADVERSE EVENTS:
Time Frame: From Day 1 up to Week 24
Description: MedDRA 24.1 coding dictionary was applied for all AE tables. The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-06946860 Q3W
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06946860 Q3W (N=10)
Anaemia (Blood and lymphatic system disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Sepsis (Infections and infestations) | 1
Transaminases increased (Investigations) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06946860 Q3W (N=10)
Anaemia (Blood and lymphatic system disorders) | 5
Monocytosis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 5
Epigastric discomfort (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Fatigue (General disorders) | 4
COVID-19 (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Oral contusion (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Electrocardiogram Q wave abnormal (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Head discomfort (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT04299048/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT04299048/SAP_001.pdf